CLINICAL TRIAL: NCT04861064
Title: Weekly Sirolimus Therapy for the Treatment of Venous and Lymphatic Malformations
Brief Title: Weekly Sirolimus Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Chelsea Shope, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00106369
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Venous Malformation; Lymphatic Malformation
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Participants will get Sirolimus (1.5-2 2mg/m2) weekly for 6 months.

SUMMARY:
In current practice, options for venous and lymphatic malformations remain limited. Recently an oral medication, sirolimus, has been found to benefit patients when taken once or twice a day for several months. Unfortunately there are many side effects associated with this medication, some of which can be severe including, neutropenia, oral ulcerations, and lab abnormalities. The purpose of this study is to determine if once weekly dosed sirolimus will be effective for the treatment of venous and lymphatic malformations. Additionally, the study will evaluate patient satisfaction and identify adverse effects. Participants will be on the medication for 6 months with an option to continue after this time period.

ELIGIBILITY:
Inclusion Criteria:

* Patient 2 years of age and older
* Venous, lymphatic, or venolymphatic malformations

Exclusion Criteria:

* Children with contraindication to use of sirolimus
* Children with history of transplant
* Children with a history of natural immunodeficiency
* Children with a history of artificially induced immunodeficiency
* Children with a history of a serious or life-threatening infection
* Children taking CYP3A4 inhibiting medications
* Children taking strong CYP3A4 inducers to avoid subtherapeutic dosing/exposure.
* Inability or unwillingness of subject or legal guardian/representative to give informed consent
* Women that are or may become pregnant o Sirolimus is a Pregnancy Category C drug. No randomized controlled studies have been done on pregnant women. Women of childbearing potential must be on effective contraception prior to, during, and for 12 weeks following sirolimus therapy.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in size of lesion | Baseline and 6 months
  Will be measuring the size of the lesions (mm) at each patient visit
Change in size of lesion through photograph | Baseline and 6 months
  Will be evaluating clinical photographs of lesions at each patient visit

SECONDARY OUTCOMES:
Number of side effects experienced | Month One
  Patient will complete side effect questionnaires at each visit
Number of side effects experienced | Month Two
  Patient will complete side effect questionnaires at each visit
Number of side effects experienced | Month Three
  Patient will complete side effect questionnaires at each visit
Number of side effects experienced | Month Four
  Patient will complete side effect questionnaires at each visit
Number of side effects experienced | Month Five
  Patient will complete side effect questionnaires at each visit
Number of side effects experienced | Month Six
  Patient will complete side effect questionnaires at each visit
Change in quality of life as assessed by questionnaire | Baseline and 6 months
  Patient will complete quality of life questionnaire at each visit
Number of participants with laboratory abnormalities | From baseline visit to 2 month visit
  Standard of care laboratory results (CBC, CMP, triglycerides) will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Shope, MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No